CLINICAL TRIAL: NCT07112261
Title: Thérapie Avatar Pour le Traitement du Trouble dépressif caractérisé réfractaire : Une étude Pilote
Brief Title: Avatar Therapy in Virtual Reality for Treatment-Resistant Major Depressive Disorder: A Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Alexandre Dumais, MD, PhD, Ciusss de L'Est de l'Île de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-3661
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Treatment-Resistant Major Depressive Disorder
Keywords: treatment-resistant major depressive disorder; relational therapy; virtual reality therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avatar Therapy (Experimental): The Avatar Intervention will take place over 10 consecutive weeks, with one session per week. Each session will last approximately 60 minutes. The goal of the intervention will be to help you reduce cravings related to your cannabis use with the use of virtual reality and avatars. The goal of the therapy is to develop strategies to improve mood and promote the fulfillment of social functioning.
  Interventions: Other: Avatar Therapy

INTERVENTIONS:
Other: Avatar Therapy — The Avatar Intervention will take place over 10 consecutive weeks, with one session per week. Each session will last approximately 60 minutes. The goal of the intervention will be to help you reduce cravings related to your cannabis use with the use of virtual reality and avatars. The goal of the therapy is to develop strategies to improve mood and promote the fulfillment of social functioning.

SUMMARY:
This pilot clinical trial aimed to evaluate the short-term efficacy of Avatar therapy for treatment-resistant major depressive disorder

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is among the most common and disabling mental health conditions worldwide. However, treatment-resistant major depressive disorder (TR-MDD) is a prevalent clinical challenge and public health concern. While various pharmacological and psychotherapeutic treatments are available, a significant proportion of individuals do not achieve adequate symptom relief. Indeed, approximately 30% to 55% of individuals with MDD remain symptomatic after two adequate antidepressant trials, and psychotherapy has shown only modest efficacy in treatment-resistant cases. In this context, our research team developed Avatar therapy, an approach using virtual reality as a therapeutic tool to treat TR-MDD. The Avatar Therapy for TR-MDD displays strong experiential and relational components that are crucially missing in conventional interventions.

Throughout the 10 therapy sessions, participants were allowed to engage in a dialogue in virtual reality with an avatar representing a person who played a significant role in their depressive symptoms, which was animated in real-time by a therapist. The primary outcomes was severity of depressive symptoms. Secondary outcomes included severity of anxiety symptoms, self-esteem, quality of life and functioning. The investigators will also explore whether the greater improvements attributable to the Avatar Therapy persist in time.

Given the high prevalence of individuals with TR-MDD and the negative repercussions for individuals, their entourage, and society, the current trial will contribute to the validation of a novel approach and create new therapeutic possibilities.

ELIGIBILITY:
Inclusion Criteria:

* Males or females over 18 years of age who meet the DSM-5 criteria for diagnosis of major depression with persistent depressive symptoms following inadequate response to two or more pharmacological treatment trials.

Exclusion Criteria:

* Current SUD for a substance
* Presence of neurological disorders ;
* Presence of a severe and unstable physical illness ;
* Inability to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms (Modified Hamilton Depression Rating Scale) | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  Depressive symptom severity was assessed using a clinician-rated scale composed of 25 items, derived from an unstructured clinical interview. Range 0-72, higher values indicating a more severe depressive symptoms.
Change in depressive symptoms (Patient Health Questionnaire-9) | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  Depressive symptom severity was also assessed using a 9-item self-report instrument. Range 0-27, higher values indicating a more severe depressive symptoms.

SECONDARY OUTCOMES:
Change in anxiety symptoms (Generalized Anxiety Disorder-7) | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  Anxiety symptom severity was assessed using a 7-item self-report questionnaire. Range 0-21, higher values indicating a more severe anxiety symptoms.
Change in self-esteem (Rosenberg Self-Esteem Scale) | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  Self-esteem was measured using a 10-item scale. Range 10-40, higher values indicate a better self-esteem,
Change in quality of life (Quality of Life Enjoyment and Satisfaction Questionnaire) | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  16-item self-reported scale measuring enjoyment and satisfaction experienced during the past week in various areas of daily functioning; Range 14-70, Higher values indicate a better satisfaction of life QLS: 21-item scale based on a semistructured interview designed to assess deficit symptoms; Range 0-126, higher values indicate a better quality of life
Deficit in functioning and disability (World Health Organization Disability Assessment Schedule 2.0) | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  Functioning and disability were assessed using a self-report instrument comprising 36 items, covering six domains: cognition, mobility, self-care, getting along with others, life activities, and participation in society. Total scores range from 36 to 180, with lower scores indicating better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Dumais, Md, PhD, Principal Investigator — University of Montreal, Centre de recherche de l'institut universitaire en santé mentale de Montréal; Stéphane Potvin, PhD, Principal Investigator — University of Montreal, Centre de recherche de l'institut universitaire en santé mentale de Montréal
Locations (1):
- Centre de recherche de l'institut universitaire en santé mentale de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No